CLINICAL TRIAL: NCT00313040
Title: Promoting Increased Physical Activity as the Main Outcome of Treatment for Overweight Persons: A Pilot Randomized Controlled Trial
Brief Title: Study to Promote Physical Activity Among Overweight Persons
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Cholestech Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79940
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Overweight; Obesity
Keywords: physical activity; sedentary; behavioral medicine; motivational interviewing
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Sedentary Behavior

INTERVENTIONS:
Behavioral: Brief Consultation with Health Counselor, workbook
Behavioral: Usual Care wait list

SUMMARY:
Recent research suggests that overweight persons who are physically active may be significantly less likely to develop health complications and less likely to die early when compared even with lean persons who are not physically active. Previous treatment programs for people who have struggled with their weight have focused almost entirely on weight loss as the main goal of treatment. Our research program has a different focus. We hope to improve health and healthy self esteem independent of body weight by focusing instead on increasing physical activity as the main goal of treatment. This is a small study designed to see if this approach would be appealing to persons who are struggling with their weight who are currently sedentary. It is designed for people who are otherwise fairly healthy for whom exercise is reasonably safe. Participants are randomly (by chance) assigned to participate in the experimental treatment program or instead to meet with their regular primary care doctor. Those who are assigned to meet with their regular doctor can access traditional weight loss resources such as Weight Watchers, Jenny Craig, Fitness centers etc... After the experiment is complete, these participants will have the opportunity to participate in the experimental treatment program.

DETAILED DESCRIPTION:
OBJECTIVE: Epidemiologic evidence suggests that overweight persons who engage in modest amounts of physical activity - even that insufficient to produce or maintain weight loss - are at significantly reduced risk for health complications including all-cause mortality. Interventions for overweight persons targeting increased physical activity rather than weight loss as the main outcome of treatment have not been well studied and could represent simpler, more sustainable, and more cost-effective approaches in addressing the obesity epidemic.

METHOD: Pilot randomized controlled trial. Sedentary patients with BMI 25-45, and no major contraindications for unsupervised physical activity recruited. Participants randomized to receive either brief consultation consisting of 3 in-person meetings, a workbook, and limited telephone contact or usual care with their medical provider including access to community weight-loss groups/resources. Intervention therapists novice pre-professional students. The intervention is manualized and coded for treatment integrity. The main outcome measures are Cohen's d effect sizes and 95% confidence intervals for the change in moderate-equivalent intensity physical activity/week at 3 months relative to baseline assessed by a blinded assessor using the Stanford 7-Day Physical Activity Recall. Secondary outcomes include effect sizes and confidence intervals for changes in cardiorespiratory fitness and depression using the modified Canadian Aerobic Fitness test and Beck Depression Inventory. Analyses to be performed by intention to treat. Missing data to be imputed by baseline observation carried forward.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-45
* not regularly physically active by staging algorithm (Norman et al,1998)
* AHA/ACSM risk class A1-A3 apparently healthy with no contraindications to medically unsupervised physical activity
* physician consent

Exclusion Criteria:

* BMI<25; BMI>45
* regularly physically active by staging algorithm (Norman et al,1998)
* AHA/ACSM risk class B or C contraindication for medically unsupervised physical activity
* physician will not consent
* diagnosis of dementia, psychotic disorder
* legal guardian or conservator appointed
* anorexia
* bulimia
* live more than one hour commute from Stanford
* no reliable means of transportation to scheduled appointments at Stanford
* unable to followup for duration of study period as result of planned move
* female and sexually active without birth control or planning to become pregnant
* unable to read and write in English
* friend or family member of enrolled participant

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Effect size and 95% CI for change in Physical Activity by 7 Day Physical Activity Recall at 3 months between groups

SECONDARY OUTCOMES:
Effect size and 95% CI for change in Cardiorespiratory Fitness at 3 months by modified Canadian Aerobic Fitness Test
Effect size and 95% CI for change in Depression by Beck Depression Inventory at 3 months
Physical Activity Staging Algorithm (Norman, 1998)
Motives for Physical Activity Measure (Ryan et al, 1997)
Self Efficacy for Overcoming Barriers to Exercise (Garcia and King, 1991)
Outcomes Expectancies for Exercise (Mascola 2004)
Health Care Climate Questionnaire (Williams, 1996)
General Causality Orientations Scale (Deci and Ryan)
Treatment Self Regulation Questionnaire (Deci and Ryan)
Mediators of Exercise Questionnaire (Mascola)
Cholestech LDX lipoprotein and glucose profile
Resting Heart Rate
Blood Pressure Omron automated sphygmomanometer
Waist Circumference
Percent Body Fat Omron bioelectric impedence
Polar OwnIndex score

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Mascola, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Result] Mascola AJ, Yiaslas TA, Meir RL, McGee SM, Downing NL, Beaver KM, Crane LB, Agras S. Framing physical activity as a distinct and uniquely valuable behavior independent of weight management: a pilot randomized controlled trial for overweight and obese sedentary persons. Eat Weight Disord. 2009 Jun-Sep;14(2-3):e148-52. doi: 10.1007/BF03327814. PMID 19934630